CLINICAL TRIAL: NCT07157826
Title: The Effect of Guided Imagery on Pain, Anxiety, Fear, Sleep Quality, Vital Signs, and Cortisol Levels in Patients Undergoing Bariatric Surgery: A Randomized Controlled Trial
Brief Title: The Effect of Guided Imagery on Bariatric Surgery Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Rumeysa Lale TORAMAN, Research Assistant, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Rumeysa TORAMAN
Record Dates: First submitted 2025-08-10; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Bariatric Surgery
Keywords: bariatric surgery; Guided Imagery; Pain; Anxiety; Fear; Cortisol
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guided Imagery Application (Experimental): On the day of hospital admission for bariatric surgery, patients in the experimental group will be administered the Personal Information Form, the Surgical Fear Questionnaire, the Richard-Campbell Sleep Questionnaire, the Visual Analog Scale (VAS) to assess pain intensity, the State-Trait Anxiety Inventory, and the parameter recording form for vital signs through face-to-face interviews conducted by the researcher. Subsequently, in line with the literature, guided imagery sessions will be implemented a total of 10 times, each lasting 10-15 minutes, as follows: morning and evening before surgery, the morning of surgery, the evening of the same day after surgery, and morning and evening on the first, second, and third postoperative days. On the morning of surgery, the Surgical Fear Questionnaire, the Richard-Campbell Sleep Questionnaire, and the State Anxiety Inventory will be administered to collect data. After the completion of the guided imagery sessions, the Surgical Fear Questionna
  Interventions: Device: Guided Imagery Application

INTERVENTIONS:
Device: Guided Imagery Application — Guided Imagery Intervention:
  Scenario-based guided imagery, one of the guided imagery techniques, will be utilized. The scenario will be developed with input from experts to promote functional recovery. Expert opinions will be obtained from a psychologist and a psychiatric nurse. The scenario will begin with breathing exercises and continue with the "safe place" technique. Patients will be instructed to listen to the audio recording using headphones in an environment free from disturbances, to set their phones to airplane mode, and to inform their relatives not to interrupt them before starting the session. Headphones will be provided by the researcher for each patient. After the content of the audio recordings is created during the initial session, it will be recorded via phone and transferred as a file to the patients' phones, with instructions on how to use it. The audio recording will last approximately 15 to 20 minutes and will include relaxing, soft background music.

SUMMARY:
The study will be conducted using a randomized controlled experimental design with experimental and control groups. Data will be collected between August 2025 and March 2026 in the General Surgery Clinic of Erzurum City Hospital. The study population will consist of patients who have undergone bariatric surgery at Erzurum City Hospital. A priori power analysis was performed to determine the sample size. According to the power analysis, based on Cohen's (Cohen, 2013) medium effect size of 0.5, with a significance level of 0.05, a 95% confidence interval, and 95% power to represent the population, it was determined that the study sample should include a total of 70 patients, with 35 patients in each group.

DETAILED DESCRIPTION:
The World Health Organization (WHO) defines obesity as an abnormal or excessive accumulation of fat in the body that may impair health. Furthermore, a body mass index (BMI) of 30 kg/m² or higher is classified as obesity, a BMI of 40 kg/m² or higher as morbid obesity, and a BMI of 50 kg/m² or higher as super obesity. Obesity is a disease with an increasing global prevalence that reduces both the quality and the length of life. Over the past 10-15 years, the rising prevalence of obesity has increased morbidity rates, adversely affected quality of life, and shortened life expectancy. This situation has turned obesity into a serious public health problem requiring urgent attention.To combat obesity, which negatively affects all body systems, methods such as medical nutrition therapy (diet), therapeutic exercise, behavioral modification therapies, and pharmacological treatments are used. In patients who do not achieve adequate results from medical and conservative approaches, surgical interventions are recommended. Influenced by social media and in pursuit of an easy and rapid solution for weight loss, obese patients often prefer surgical methods (bariatric surgery). The lack of guidance from healthcare teams regarding surgery and insufficient therapeutic communication with patients can lead to anxiety and depression during hospitalization. Pharmacological and non-pharmacological approaches can prevent disease- and surgery-related symptoms, reduce anxiety, and contribute to improved sleep quality. These methods provide emotional, mental, social, and behavioral benefits to patients. Techniques such as hypnosis, biofeedback, meditation, and imagery enhance the interaction between the body and mind, thereby promoting healing. These practices activate the body's self-healing potential by influencing the mind. Guided imagery allows patients to feel happy, comfortable, peaceful, and safe, and to develop positive thoughts. It can be applied with soft background music to facilitate relaxation and help patients distance themselves from negative thoughts. Guided imagery is a mind-body intervention that uses the patient's imagination and mental processes to create a mental representation of an object, place, event, or situation perceived through the senses. It is considered a relaxation technique focusing on the interaction between the brain, mind, body, and behavior. Patients are instructed to focus on pleasant images that replace negative or stressful emotions. Guided imagery can be self-directed, facilitated by a professional, or delivered through a recording.This study was planned considering the need for evidence on the use of guided imagery in preoperative and postoperative care in the context of nursing practice. Given the mind-body connection between preoperative anxiety and major elective surgical procedures, it is hypothesized that guided imagery may be effective in reducing pain, anxiety, fear, and improving sleep quality, cortisol levels, blood glucose, and vital signs in patients undergoing bariatric surgery before and after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study
* Ability to communicate verbally
* No history of psychiatric disorders
* Undergoing laparoscopic bariatric surgery using the Sleeve Gastrectomy method
* Ability to use a smartphone
* No prior experience with guided imagery intervention

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | up to 24 hours
  The Personal Information Form, developed by the researcher based on a review of the relevant literature, consists of a total of 16 questions. It includes items related to gender, age, education level, marital status, and previous surgical history.
The Surgical Fear Scale | up to 24 hours
  Developed by Theunissen et al. in 2014 to assess the fear levels of patients scheduled for surgical procedures, this 8-item Likert-type scale evaluates short-term surgical fears with items 1-4 and long-term surgical fears with items 5-8. Each item is scored on a scale from 0 ("not afraid at all") to 10 ("very afraid"), resulting in a total score ranging from 0 to 80. Higher scores indicate greater levels of surgical fear (Theunissen et al., 2014). The Turkish validity and reliability study conducted by Bağdigen and Özlü (2018) reported a Cronbach's alpha coefficient of 0.93.
Richard-Campbell Sleep Questionnaire | up to 24 hours
  The Richard-Campbell Sleep Questionnaire was developed by Richards in 1987 and its Turkish validity and reliability study was conducted by Özlü and Özer in 2015 . The scale consists of 6 items that assess various aspects of nighttime sleep, including sleep depth, sleep latency, frequency of awakenings, duration of awakening after sleep onset, sleep quality, and noise level in the environment. Each item is scored on a scale from 0 to 100. However, when calculating the total score, the 6th item (noise level) is excluded, and the evaluation is based on the first 5 items. Higher scores indicate better sleep quality. The total score is obtained by dividing the sum of the item scores by the number of items. Scores ranging from 0 to 25 indicate very poor sleep quality, while scores between 76 and 100 indicate very good sleep quality.
Visual Analog Scale for Pain (VAS) | up to 24 hours
  Developed by Price et al. (1983), this scale measures the intensity of pain using a 10 cm vertical or horizontal line with endpoints labeled as "no pain" (0) and "worst possible pain" (10). The patient marks a point corresponding to their perceived pain intensity, and the distance from the "no pain" end to the marked point is measured in centimeters, representing the pain score. Higher scores indicate greater pain intensity.
State-Trait Anxiety İnventory (STAI-I, STAI-II) | up to 24 hours
  It is a test developed by Spielberger et al. that measures state and trait anxiety levels. Its validity and reliability in Turkey was done by Oner and Le Compte. The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings, and the 20-item 'trait anxiety scale', which was created to determine the feelings in general. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
Parameter Tracking Form | up to 24 hours
  Before and after bariatric surgery, patients' heart rate, blood pressure, and oxygen saturation will be measured and recorded in this form. In addition, to assess stress levels, blood cortisol measurements will be performed. Blood samples for cortisol will be collected in the morning (between 07:30-08:30) in appropriate tubes, promptly transported to the laboratory, and analyzed under cold chain conditions. Serum or plasma will be separated and analyzed using standard devices. All procedures will be carried out in the Erzurum City Hospital laboratory according to existing standard protocols and high-quality criteria, and results will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: RUMEYSA LALE TORAMAN, Principal Investigator — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No